CLINICAL TRIAL: NCT05262894
Title: Evaluation of Gas Propagation in Snow During Breathing of Subjects Under Simulated Avalanche Snow
Acronym: GasProp
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Czech Technical University in Prague (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 2022-Bradler
Record Dates: First submitted 2022-02-21; First posted 2022-03-02 (Actual); Last update posted 2022-03-02 (Actual); Status verified 2022-02

CONDITIONS: Accident Caused by Snow Avalanche
Keywords: snow; avalanche; hypercapnia; diffusion
MeSH Terms: conditions — Hypercapnia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Breathing in the snow (Experimental): Breathing in the snow using a specially designed apparatus and measuring the respiratory gases distribution in snow.
  Interventions: Other: extreme hypercapnia induced by ventilation insufficiency

INTERVENTIONS:
Other: extreme hypercapnia induced by ventilation insufficiency — Re-breathing of gas by breathing into the simulated avalanche snow

SUMMARY:
The study is aimed at investigation of respiratory gases propagation in snow. The study involves volunteers breathing into the snow whereas concentrations of gases are measured at various positions in the snow.

DETAILED DESCRIPTION:
The study is aimed at investigation of respiratory gases (oxygen and carbon dioxide) propagation in the simulated avalanche snow. The study involves volunteers breathing into the snow whereas concentrations of gases are measured at various positions in the snow. A special apparatus was created for sampling and measurement of gas concentrations and to assure stable geometry of the experiment required for data evaluation.

ELIGIBILITY:
Inclusion Criteria:

* healthy and fit volunteers, classified as The American Society of Anesthesiologists class I
* without a smoking history

Exclusion Criteria:

* Tiffeneau Index less than 0.70
* any cardiovascular or respiratory condition

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 50 (Estimated)
Dates: Start 2022-02-07 (Actual); Primary Completion 2025-05-31 (Estimated); Study Completion 2025-05-31 (Estimated)

PRIMARY OUTCOMES:
The length of breathing | Continuously within up to 20 minute interval from the beginning of the breathing experiment
  Time to termination of the breathing experiment due to the decision of the tested subject, or determined by high end-tidal carbon dioxide value or by the order by the clinician assessing the health status of the subjects.

CONTACTS AND LOCATIONS:
Overall Officials: Karel Roubik, prof., Principal Investigator — Czech Technical University in Prague, Fac. of Biomedical Engineering
Locations (1):
- Czech Technical University, Faculty of Biomedical Engineering, Kladno, Czechia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Roubik K, Sieger L, Sykora K. Work of Breathing into Snow in the Presence versus Absence of an Artificial Air Pocket Affects Hypoxia and Hypercapnia of a Victim Covered with Avalanche Snow: A Randomized Double Blind Crossover Study. PLoS One. 2015 Dec 14;10(12):e0144332. doi: 10.1371/journal.pone.0144332. eCollection 2015. PMID 26666523
- [Background] Roubik K, Sykora K, Sieger L, Ort V, Horakova L, Walzel S. Perlite is a suitable model material for experiments investigating breathing in high density snow. Sci Rep. 2022 Feb 8;12(1):2070. doi: 10.1038/s41598-022-06015-y. PMID 35136116